CLINICAL TRIAL: NCT02667535
Title: Pharmacokinetics, Pharmacodynamics and Safety Comparative Trial of Isosorbide Mononitrate Gel in Participants With Anal Fissure and Healthy Volunteers.
Brief Title: PK, PD and Safety Comparative Trial of Isosorbide Mononitrate Gel in Healthy Participants and With Anal Fissure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been cancelled and it has not been initiated.
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDN 001/16
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Anal Fissure
MeSH Terms: conditions — Fissure in Ano | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Isosorbide Mononitrate 2.0% healthy (Experimental): Isosorbide Mononitrate gel 2.0% - 2g Anorectal usage Once daily Healthy volunteers
  Interventions: Drug: Isosorbide Mononitrate
- Isosorbide Mononitrate 0.5% anal fissure (Experimental): Isosorbide Mononitrate gel 0.5% - 2g Anorectal usage Once daily Participants with anal fissure
  Interventions: Drug: Isosorbide Mononitrate
- Isosorbide Mononitrate 1.0% anal fissure (Experimental): Isosorbide Mononitrate gel 1.0% - 2g Anorectal usage Once daily Participants with anal fissure
  Interventions: Drug: Isosorbide Mononitrate
- Isosorbide Mononitrate 2.0% anal fissure (Experimental): Isosorbide Mononitrate gel 2.0% - 2g Anorectal usage Once daily Participants with anal fissure
  Interventions: Drug: Isosorbide Mononitrate

INTERVENTIONS:
Drug: Isosorbide Mononitrate — Healthy volunteers will receive 2g (2.0%) of investigational product at a single dose, and will undergo a washout period of 7 days; subsequently, they will receive 2g of investigational product once daily, for 7 consecutive days.
  Participants with anal fissure will receive 2g of investigational product, either at 0.5%, 1.0% or 2.0%, at a single dose, and will undergo a washout period of 7 days; subsequently, they will receive 2g of investigational product, either at 0.5%, 1.0% or 2.0%, once daily, for 7 consecutive days.

SUMMARY:
This is a Phase I trial to evaluate Pharmacokinetics, Pharmacodynamics and Safety of Isosorbide Mononitrate gel for usage in participants with anal fissure and healthy volunteers. Three doses will be used in patients with anal fissure (0.5%, 1.0% or 2.0%) and healthy volunteers will receive 2.0% dose. All treatment will last 7 days.

DETAILED DESCRIPTION:
This is a Phase I, open-label, parallel trial to evaluate Pharmacokinetics, Pharmacodynamics and Safety of Isosorbide Mononitrate gel for usage in participants with anal fissure and healthy volunteers.

Investigational product will be randomly assigned as follows:

* healthy volunteers will receive 2g (2.0%) of investigational product at a single dose, and will undergo a washout period of 7 days; subsequently, they will receive 2g of investigational product once daily, for 7 consecutive days;
* participants with anal fissure will receive 2g of investigational product, either at 0.5%, 1.0% or 2.0%, at a single dose, and will undergo a washout period of 7 days; subsequently, they will receive 2g of investigational product, either at 0.5%, 1.0% or 2.0%, once daily, for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18 years-old;
* Body mass index (BMI) ≥ 19 Kg/m2 and ≤ 35 Kg/m2;
* For healthy volunteers: good health conditions or without significant diseases, according to best medical judgement, according to protocol requirements and study evaluations: medical history, blood pressure and heart rate measurements, physical examination, electrocardiogram (ECG) and screening laboratory tests;
* For participants with the condition under study: anal fissure;
* Ability to understand the nature and objectives of the trial, including risks and adverse events; willingness to cooperate with the researcher and proceed according to all study requirements, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Known hypersensitivity to the investigational products (naproxen or rebamipide) or chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug;
* Chronic therapy with any drugs, except oral contraceptives and medication authorized by principal investigator (each case to be individually evaluated);
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic or psychiatric disease; hypotension or hypertension, or any other co-morbidity that requires priority immediate treatment ot that, at principal investigator discretion, might interfere with study participation or expose study participant to risks other than predicted;
* Deviations on screening laboratory results that are considered as clinically relevant by the principal investigator;
* Smoking;
* History of drugs and alcohol addiction or excessive alcohol consumption (> 35 g/ day);
* Use of regular medications within 2 weeks prior study enrollment or use of any medications within one week prior to study enrollment, except oral contraceptives or cases which, based on drug's or metabolite's half-life, complete elimination can be assumed;
* Treatment, within 6 months before the trial, with any drugs known to have a well established toxic potential to major organs;
* Participation in any other experimental research or administration of any experimental drug within six months before this trial;
* Donation or loss of 450 mL of blood (or more) within 3 months before the trial, or 4 donations within 12 months before the trial;
* Any condition, according to investigator's best judgement, that prevents the subject to participate in the trial;
* Pregnancy, labor or miscarriage with 12 weeks before admission predicted date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics, area under the curve time zero - last (AUC t0-last) | 7 days
Pharmacokinetics, area under the curve time zero - infinite (AUC t0-inf) | 7 days
Pharmacokinetics, constant of elimination (Ke) | 7 days
Pharmacokinetics, half-life (t1/2) | 7 days

SECONDARY OUTCOMES:
Safety, by number of adverse events | 7 days
Safety, by blood pressure measurement | 7 days
Anorectal muscle contractility, by anorectal manometry | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas

IPD SHARING:
Plan to Share IPD: No